CLINICAL TRIAL: NCT03955393
Title: THE ROLE OF 18F-FAZA PET IMAGING TECHNIQUE IN DETECTING LYMPH NODE METASTASES IN RENAL CELL CARCINOMA PATIENTS
Brief Title: FAZA PET IMAGING IN DETECTING LYMPH NODE METASTASES IN RENAL CELL CARCINOMA PATIENTS
Acronym: FAZA
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Umberto Capitanio, Principal Investigator, IRCCS San Raffaele
Other Study IDs: FAZA RCC LNI
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: LYMPH NODE METASTASES; 18F-FAZA PET IMAGING TECHNIQUE
MeSH Terms: conditions — Carcinoma, Renal Cell; Lymphatic Metastasis | interventions — fluoroazomycin arabinoside

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LYMPH NODE METASTASES IN RENAL CELL CARCINOMA PATIENTS: Twenty patients candidates to radical nephrectomy and extended lymphadenectomy for clinical T4 cancers (clinical Nany) or renal masses with evidence of lymphadenopathies at preoperative CT scan (clinical Tany N1) or larger tumor (clinical Tany Nany and max diameter>10 cm). RCC candidates to surgery will receive a single intravenous infusion of 18F-FAZA. Surgery will be scheduled within 1 week after infusion. PET and CT scanning of the abdomen will be planned before surgery.
  Interventions: Other: 18F-FAZA PET IMAGING TECHNIQUE IN DETECTING LYMPH NODE METASTASES IN RENAL CELL CARCINOMA PATIENTS

INTERVENTIONS:
Other: 18F-FAZA PET IMAGING TECHNIQUE IN DETECTING LYMPH NODE METASTASES IN RENAL CELL CARCINOMA PATIENTS — 18F-FAZA is a highly selective PET radiotracer of hypoxia, which has been recently developed and tested in several studies (10-14). 18F-FAZA has been demonstrated to be a marker of hypoxia and pathological metabolic patterns which are common to all renal cancers.
  Other Names: 18F-FAZA

SUMMARY:
In renal cell carcinoma (RCC) patients, lymph node metastases detection and treatment are the most critical issues in daily clinical decision-making. Indeed, conversely to other oncological settings, a) nodal status imaging, b) sentinel node technique and c) standard lymphadenectomy have been demonstrated inadequate in the staging and management of RCC patients. A novel, accurate, standardized imaging technique is urgently needed in RCC setting to detect macro and micro nodal invasion, to identify those patients who are at higher risk of having nodal metastases, to accurately plan the best management. Recent studies suggested combining 18F-FAZA PET with CT scanning in the detection of cancer-induced hypoxia.The investigators propose to test 18F-FAZA PET-CT in detecting nodal metastases to improve the management of RCC patients.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 18 years with diagnosis of RCC;
* patients candidates to radical nephrectomy and extended lymphadenectomy
* clinical T4 cancers or renal masses with evidence of lymphadenopathies at preoperative CT scan or larger tumor (max diameter>10 cm)
* performance status 0-1;
* expected survival time of at least 3 months;
* recovery from toxic effects of any previous treatment;
* serum biochemical and haematological measurements within healthy parameters.
* Female patients of childbearing age were requested to have a negative pregnancy test
* ability to understand and understand informed consent
* acceptance and signature of informed consent

Exclusion Criteria:

* other medical conditions that might limit the amount of antibody to be administered;
* New York Heart Association Class III/IV cardiac disease;
* pregnancy and breastfeeding
* eGFR<30;
* women of child-bearing age who do not agree to use contraceptives to avoid pregnancy;
* history of autoimmune hepatitis;
* allergy to iodine;
* unavailability or immunological and clinical follow-up assessments;
* participation in another clinical trial involving an investigational agent within 4 weeks of study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients candidates to radical nephrectomy and extended lymphadenectomy for clinical T4 cancers (clinical Nany) or renal masses with evidence of lymphadenopathies at preoperative CT scan (clinical Tany N1) or larger tumor (clinical Tany Nany and max diameter>10 cm).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Test the performance of 18F-FAZA | 120 minutes
  To test the performance of 18F-FAZA PET technique in detecting nodal metastases in RCC patients

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ljungberg B, Cowan NC, Hanbury DC, Hora M, Kuczyk MA, Merseburger AS, Patard JJ, Mulders PF, Sinescu IC; European Association of Urology Guideline Group. EAU guidelines on renal cell carcinoma: the 2010 update. Eur Urol. 2010 Sep;58(3):398-406. doi: 10.1016/j.eururo.2010.06.032. Epub 2010 Jul 12. PMID 20633979
- [Background] Capitanio U, Becker F, Blute ML, Mulders P, Patard JJ, Russo P, Studer UE, Van Poppel H. Lymph node dissection in renal cell carcinoma. Eur Urol. 2011 Dec;60(6):1212-20. doi: 10.1016/j.eururo.2011.09.003. Epub 2011 Sep 13. PMID 21940096
- [Background] Studer UE, Scherz S, Scheidegger J, Kraft R, Sonntag R, Ackermann D, Zingg EJ. Enlargement of regional lymph nodes in renal cell carcinoma is often not due to metastases. J Urol. 1990 Aug;144(2 Pt 1):243-5. doi: 10.1016/s0022-5347(17)39422-3. PMID 2374186
- [Background] Lughezzani G, Capitanio U, Jeldres C, Isbarn H, Shariat SF, Arjane P, Widmer H, Perrotte P, Montorsi F, Karakiewicz PI. Prognostic significance of lymph node invasion in patients with metastatic renal cell carcinoma: a population-based perspective. Cancer. 2009 Dec 15;115(24):5680-7. doi: 10.1002/cncr.24682. PMID 19824083
- [Background] Vasselli JR, Yang JC, Linehan WM, White DE, Rosenberg SA, Walther MM. Lack of retroperitoneal lymphadenopathy predicts survival of patients with metastatic renal cell carcinoma. J Urol. 2001 Jul;166(1):68-72. PMID 11435825
- [Background] Stenzl A, Cowan NC, De Santis M, Jakse G, Kuczyk MA, Merseburger AS, Ribal MJ, Sherif A, Witjes JA. The updated EAU guidelines on muscle-invasive and metastatic bladder cancer. Eur Urol. 2009 Apr;55(4):815-25. doi: 10.1016/j.eururo.2009.01.002. Epub 2009 Jan 13. PMID 19157687
- [Background] Heidenreich A, Bellmunt J, Bolla M, Joniau S, Mason M, Matveev V, Mottet N, Schmid HP, van der Kwast T, Wiegel T, Zattoni F; European Association of Urology. EAU guidelines on prostate cancer. Part 1: screening, diagnosis, and treatment of clinically localised disease. Eur Urol. 2011 Jan;59(1):61-71. doi: 10.1016/j.eururo.2010.10.039. Epub 2010 Oct 28. PMID 21056534
- [Background] Blom JH, van Poppel H, Marechal JM, Jacqmin D, Schroder FH, de Prijck L, Sylvester R; EORTC Genitourinary Tract Cancer Group. Radical nephrectomy with and without lymph-node dissection: final results of European Organization for Research and Treatment of Cancer (EORTC) randomized phase 3 trial 30881. Eur Urol. 2009 Jan;55(1):28-34. doi: 10.1016/j.eururo.2008.09.052. Epub 2008 Oct 1. PMID 18848382
- [Background] Beyer T, Czernin J, Freudenberg LS. Variations in clinical PET/CT operations: results of an international survey of active PET/CT users. J Nucl Med. 2011 Feb;52(2):303-10. doi: 10.2967/jnumed.110.079624. Epub 2011 Jan 13. PMID 21233186
- [Background] Studer UE, Birkhauser FD. Lymphadenectomy combined with radical nephrectomy: to do or not to do? Eur Urol. 2009 Jan;55(1):35-7. doi: 10.1016/j.eururo.2008.09.056. Epub 2008 Oct 7. No abstract available. PMID 18848383
- [Background] Capitanio U, Pepe G, Incerti E, Larcher A, Trevisani F, Luciano R, Mapelli P, Bettinardi V, Monterisi C, Necchi A, Cascinu S, Bernardi R, Bertini R, Doglioni C, Gianolli L, Salonia A, Picchio M, Montorsi F. The role of 18F-FAZA PET/CT in detecting lymph node metastases in renal cell carcinoma patients: a prospective pilot trial. Eur J Nucl Med Mol Imaging. 2021 Feb;48(2):554-560. doi: 10.1007/s00259-020-04936-2. Epub 2020 Jul 8. PMID 32638098